CLINICAL TRIAL: NCT05068778
Title: Development of an Artificial Intelligence Platform / Digital Dental Hygienist to Improve Compliance in Periodontal Maintenance Patients
Brief Title: Development of an AI App to Improve Compliance in Periodontal Maintenance Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McGuire Institute (Industry)
Collaborators: Asua, Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: Asua 001-2020
Record Dates: First submitted 2021-08-27; First posted 2021-10-06 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Artificial Intelligence Application — AI application through smart phone

SUMMARY:
An Artificial Intelligence platform to develop an app which improves compliance in periodontal treatments

DETAILED DESCRIPTION:
To develop the accuracy of an AI-determined decision-making process for compliance score (CS) assignment, to assess clinical efficacy, and develop patient reported outcomes of AI-facilitated communication / education on a subject's oral health behaviors over successive maintenance visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 to 75-yrs of age
2. Subjects with diagnosis and treatment of Generalized and/or Localized Periodontitis Stages I, II, or III; grades A-C and or Peri-implantitis (Generalized Mild, Moderate, or Advanced Chronic Periodontitis) who are following a periodontal maintenance interval of every three months.
3. Subjects are able to provide self-care (oral hygiene) without disabilities requiring assistance with daily oral hygiene measures.
4. Subjects will have read, understood and signed an institutional review board (IRB) approved Informed Consent Form (ICF).
5. Subjects must be able and willing to follow study procedures and instructions.

Exclusion Criteria:

1. Subjects who do not own or are incapable of interacting with a smart phone or device
2. Subjects who are incapable of operating an application on a smart phone or device
3. Subjects who are not compliant with periodontal maintenance / recall intervals (Based on Wilson's classification as any lack of compliance with their recommended maintenance interval- therefore exclude subjects who demonstrate erratic compliance or noncompliance)18
4. Subjects who require active periodontal therapy during the study
5. Subjects who are on immunosuppressive medications, chemotherapy, or radiation therapy which would adversely affect their periodontal stability.
6. Subjects participating in other clinical studies involving therapeutic intervention (either medical or dental).
7. Subjects, who in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

   -

   Exclusion Criteria:

   -

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 50 subjects minimum, 18-75 years of age, treated for periodontitis in a private practice who are currently following a periodontal maintenance regimen.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
To identify the input variables the AI utilizes to arrive at CS assignment and message selection for subject interaction via DDH app | through study completion, approximately 7 months
  Digital hygiene app will provide messages to subjects via their smartphone regarding their their lst maintenance appointment and throughout the study.

SECONDARY OUTCOMES:
Compliance Score Accuracy | 6 months
  the increase the compliance score ant 3 and 6 months after subject begins use of the AI app
change in recession | 6 months
  number of subjects with a lesser degree of recession from baseline to end of study due to increased subject compliance
change in probing depth | 6 months
  number of subjects with a lesser probing depth from baseline to end of study due to increased subject compliance
change in clinical attachment level | 6 months
  number of subjects with improved clinical attachment level due to increased subject compliance
change in gingival inflammation | 6 months
  number of subjects with a reduction in gingival inflammation due to increased subject compliance
decrease mobility | 6 months
  number of subjects showing a decreased degree of tooth mobility due to increased subject compliance

OTHER OUTCOMES:
PRO | 6 months
  PRO for subject experience using the AI app system
Subject demographics | 6 months
  determination of demographics on subjects with periodontal disease
AI generated surveys | 6 months
  survey to determine subjects progress, risk disease, oral hygiene needs, coping and goal setting abilities, and compliance
Hygienist In office subject survey | 6 months
  to measure subjects hygiene and other life events (e.g. work stress)

CONTACTS AND LOCATIONS:
Overall Officials: Rick Heard, DDS, Study Director — The McGuire Institute
Locations (2):
- United States (2):
  - Metro West Orthodontics & Periodontics, La Vista, Nebraska
  - Perio Health Professionals, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shapiro SC. Encyclopedia of Artificial Intelligence. New York: Wiley; 1992.
- [Background] Park WJ, Park JB. History and application of artificial neural networks in dentistry. Eur J Dent. 2018 Oct-Dec;12(4):594-601. doi: 10.4103/ejd.ejd_325_18. PMID 30369809
- [Background] Jackson P. Introduction to Expert Systems. London: Addison Wesley; 1986
- [Background] Khanna S. Artificial intelligence: contemporary applications and future compass. Int Dent J. 2010 Aug;60(4):269-72. PMID 20949757
- [Background] Xie X, Wang L, Wang A. Artificial neural network modeling for deciding if extractions are necessary prior to orthodontic treatment. Angle Orthod. 2010 Mar;80(2):262-6. doi: 10.2319/111608-588.1. PMID 19905850
- [Background] Kim EY, Lim KO, Rhee HS. Predictive modeling of dental pain using neural network. Stud Health Technol Inform. 2009;146:745-6. PMID 19592958
- [Background] Reddy MS, Shetty SR, Shetty RM, Vannala V, Sk S. Future of periodontics lies in artificial intelligence: Myth or reality? J Investig Clin Dent. 2019 Nov;10(4):e12423. doi: 10.1111/jicd.12423. Epub 2019 May 23. No abstract available. PMID 31120578
- [Background] Wilson TG Jr, Glover ME, Malik AK, Schoen JA, Dorsett D. Tooth loss in maintenance patients in a private periodontal practice. J Periodontol. 1987 Apr;58(4):231-5. doi: 10.1902/jop.1987.58.4.231. PMID 3295181
- [Background] Miyamoto T, Kumagai T, Jones JA, Van Dyke TE, Nunn ME. Compliance as a prognostic indicator: retrospective study of 505 patients treated and maintained for 15 years. J Periodontol. 2006 Feb;77(2):223-32. doi: 10.1902/jop.2006.040349. PMID 16460248
- [Background] McGuire MK, Nunn ME. Prognosis versus actual outcome. III. The effectiveness of clinical parameters in accurately predicting tooth survival. J Periodontol. 1996 Jul;67(7):666-74. doi: 10.1902/jop.1996.67.7.666. PMID 8832477
- [Background] Needleman I, Nibali L, Di Iorio A. Professional mechanical plaque removal for prevention of periodontal diseases in adults--systematic review update. J Clin Periodontol. 2015 Apr;42 Suppl 16:S12-35. doi: 10.1111/jcpe.12341. PMID 25495962
- [Background] Tonetti MS, Eickholz P, Loos BG, Papapanou P, van der Velden U, Armitage G, Bouchard P, Deinzer R, Dietrich T, Hughes F, Kocher T, Lang NP, Lopez R, Needleman I, Newton T, Nibali L, Pretzl B, Ramseier C, Sanz-Sanchez I, Schlagenhauf U, Suvan JE. Principles in prevention of periodontal diseases: Consensus report of group 1 of the 11th European Workshop on Periodontology on effective prevention of periodontal and peri-implant diseases. J Clin Periodontol. 2015 Apr;42 Suppl 16:S5-11. doi: 10.1111/jcpe.12368. PMID 25639948
- [Background] Asimakopoulou K, Nolan M, McCarthy C, Newton JT. The effect of risk communication on periodontal treatment outcomes: A randomized controlled trial. J Periodontol. 2019 Sep;90(9):948-956. doi: 10.1002/JPER.18-0385. Epub 2019 Apr 17. PMID 30997690
- [Background] Amerio E, Mainas G, Petrova D, Giner Tarrida L, Nart J, Monje A. Compliance with supportive periodontal/peri-implant therapy: A systematic review. J Clin Periodontol. 2020 Jan;47(1):81-100. doi: 10.1111/jcpe.13204. Epub 2019 Nov 13. PMID 31562778
- [Background] Asimakopoulou K, Newton JT, Daly B, Kutzer Y, Ide M. The effects of providing periodontal disease risk information on psychological outcomes - a randomized controlled trial. J Clin Periodontol. 2015 Apr;42(4):350-5. doi: 10.1111/jcpe.12377. Epub 2015 Mar 24. PMID 25682859
- [Background] Newton JT, Asimakopoulou K. Managing oral hygiene as a risk factor for periodontal disease: a systematic review of psychological approaches to behaviour change for improved plaque control in periodontal management. J Clin Periodontol. 2015 Apr;42 Suppl 16:S36-46. doi: 10.1111/jcpe.12356. PMID 25639708
- [Background] Free C, Knight R, Robertson S, Whittaker R, Edwards P, Zhou W, Rodgers A, Cairns J, Kenward MG, Roberts I. Smoking cessation support delivered via mobile phone text messaging (txt2stop): a single-blind, randomised trial. Lancet. 2011 Jul 2;378(9785):49-55. doi: 10.1016/S0140-6736(11)60701-0. PMID 21722952
- [Background] Wilson TG Jr, Glover ME, Schoen J, Baus C, Jacobs T. Compliance with maintenance therapy in a private periodontal practice. J Periodontol. 1984 Aug;55(8):468-73. doi: 10.1902/jop.1984.55.8.468. PMID 6384465
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Background] Miller SC. Textbook of Periodontia: Philadelphia, Blakiston; 1938
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182